CLINICAL TRIAL: NCT06921369
Title: The Effect of Compassionate Care Training Given According to Watson's Human Caring Model on Nurses' Compassion Levels and Caring Behaviors
Brief Title: The Effect of Compassionate Care Education on Nurses
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kırıkkale University (Other)
Responsible Party: Principal Investigator, Gönül GÜMÜŞ, Lecturer (MSc), Kırıkkale University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 04-371
Record Dates: First submitted 2025-03-18; First posted 2025-04-10 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Nursing; Compassion
Keywords: nursing; compassionate care; Video-assisted teaching; Caring behaviors

STUDY DESIGN:
Intervention Model Description: Single-group pre-test-post-test quasi-experimental study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Group Assignment (Experimental): Nurse group
  Interventions: Other: Compassion Competence Scale; Other: Caring Behaviors Scale; Other: Nurse Feedback Form on Compassionate Care Training

INTERVENTIONS:
Other: Compassion Competence Scale — Compassion Competence Scale
Other: Caring Behaviors Scale — Caring Behaviors Scale
Other: Nurse Feedback Form on Compassionate Care Training — Nurse Feedback Form on Compassionate Care Training

SUMMARY:
Compassion is an important concept underlying relationships between people. Compassion is a complex, multifaceted psychological and social process. Professional values form the basis of nursing care. The concept of compassion is one of these professional values, as well as one of the essential components of care that facilitates nursing care. Compassion-based care provides patient-centered care with a holistic approach while increasing the quality of care. Despite this importance, many healthcare professionals remain inadequate regarding compassionate care. The idea that compassion is innate or learned in people causes various difficulties in teaching compassion. Compassionate care is an emotion that can be taught and developed with innovative interactive methods along with developing technology. Methods such as video-supported teaching and case analysis, which are widely used in nursing education, contribute to developing cognitive and affective skills such as interpretation, critical thinking, and problem-solving in nurses. In this context, it is aimed to implement compassionate care training, developed based on Watson's Human Caring Model, on nurses by enriching it with video-supported teaching and case analysis methods, and to evaluate the effect of this training on nurses' compassion levels and caring behaviors.

DETAILED DESCRIPTION:
The research will be conducted as a single group pre-test-post-test quasi-experimental study to determine the effect of compassionate care training, which will be given using video-assisted teaching and case analysis methods according to Watson's Human Caring Model, on nurses' compassion levels and caring behaviors.

The universe of the research will consist of 220 nurses working in the Surgery Clinic, Internal Medicine Clinic, Intensive Care Unit and Emergency Department at Kırıkkale University Faculty of Medicine Hospital between 20.12.2025 and 20.02.2026. The power of the study was measured with the G*Power 3.1.9.2 package program. The sample size was calculated with a medium effect width. Accordingly, the minimum sample size to be studied for 95% power at a significance level of 0.05 and an effect width of 0.5 was predicted to be 54. The research aims to reach 60 people, considering the losses.

The sample will consist of nurses who meet the research criteria, are not on leave during the research period, and agree to participate in the research.

Implementation of the Research:

Preparation phase:

"Preparation of the Content of the Compassionate Care Education Program to be Given According to Watson's Human Care Model" Compassionate care training for nurses, based on Watson's Human Caring Model, has been developed in accordance with literature. The training is planned in four sessions. In sessions 2, 3, and 4, videos from the prepared scenarios will be shown, and case studies will be conducted with the nurses (six case scenarios containing compassionate care behaviors and six scenarios containing negative versions of the same scenario without compassionate care behaviors, for a total of 12 scenarios).

Implementation of the Study During the implementation phase of the study, pre-tests will be conducted between December 20, 2025, and February 20, 2026, by asking all nurses, for whom written consent has been obtained, to complete the "Descriptive Characteristics Form," the "Compassion Competence Scale," and the "Caring Behaviors Scale." All nurses in the sample group will receive compassionate care training implemented according to Watson's Human Caring Model. During the second, third, and fourth sessions of the training, videos taken from the prepared scenarios will be watched, and case studies will be conducted with the nurses. Following this four-week training program, post-test measurements will be taken by asking them to complete the "Compassion Competence Scale" and the "Caring Behaviors Scale." After the compassionate care training implemented according to Watson's Human Caring Model, the "Compassion Competence Scale" and "Caring Behaviors Scale" measurements will be repeated at the end of the first and second months. The training will be delivered in groups of 12 nurses, depending on their work schedules. Nurses will be divided into groups of 12, and the same training session will be delivered face-to-face to five different groups on different days that week, outside of working hours, at the nurses' convenience, in a meeting room at the hospital. After the training, nurses will be asked to complete a "Nurse Feedback Form on Compassionate Care Training."

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study,
* Understanding and using Turkish effectively,
* Not being on leave during the study.

Exclusion Criteria:

* Nurses who answered the data collection forms incompletely,
* Nurses who did not want to continue the study,
* Nurses who did not participate in even one of the compassionate care education programs of the study.

Max Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2026-01-16 (Estimated); Study Completion 2026-02-20 (Estimated)

PRIMARY OUTCOMES:
Compassion Competence Scale | 12 weeks from enrollment to the end of training
  "Compassion Competence Scale"; consists of 3 sub-dimensions: "Communication," which expresses understanding and compassion towards patients and their families; "Sensitivity," which expresses the ability to notice and respond to changes in patients' emotions through careful observation; and "Insight," which expresses the ability to clearly understand patients and comprehensively meet their needs and conditions based on professional knowledge. The scale is a 5-point Likert-type scale with 11 items. The scale is interpreted by calculating the mean scores of the items. The highest score that can be obtained from the scale is 5, and the lowest score is 1. As the score increases, the level of compassion competence increases.

SECONDARY OUTCOMES:
Caring Behaviors Scale | 12 weeks from enrollment to the end of training
  The original version of the Caring Behaviors Scale consists of 42 items. The Turkish version has 30 items and is divided into three subscales: "respect for others" (items 1-10), "professional knowledge and attitude" (items 11-20), and "being available to the individual" (items 21-30). The scale is scored using a six-point Likert-type rating system ranging from "never" to "always" and does not include reverse items. The total score ranges from 30 to 180, with no specified cutoff point. High scores indicate a positive perception of nursing care, while low scores indicate a weak perception.with the Compassionate Care Checklist will be prepared in a table form with the expressions "Strongly Disagree," "Disagree," "Undecided," "Agree," and "Strongly Agree." In the scoring, the expression "Strongly Disagree" will be given 1 point, "Disagree" 2 points, "Undecided" 3 points, "Agree" 4 points, and "Strongly Agree" 5 points. . As the score increases, compassionate care attitudes increases.
Nurse Feedback Form on Compassionate Care Training | 12 weeks from enrollment to the end of training
  This is a form created by the researcher with open-ended questions to obtain nurses' opinions on compassionate care education according to Watson's Human Caring Model. The form includes three open-ended questions that question nurses' feelings and thoughts about the content of the education and the methods used in the education.

CONTACTS AND LOCATIONS:
Overall Officials: Gönül GÜMÜŞ, Principal Investigator — Kırıkkale University
Locations (1):
- Kirikkale University, Kırıkkale, Kırıkkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It will not be shared because it is not ethically appropriate.

REFERENCES:
- [Background] Abate M, Tadesse N, Mitiku K. Level of compassionate health care service provision and its associated factors among health professionals working in public hospitals of Addis Ababa: health professionals' perspective. Heliyon. 2022 Mar 23;8(3):e09160. doi: 10.1016/j.heliyon.2022.e09160. eCollection 2022 Mar. PMID 35846442
- [Background] Adam D, Taylor R. Compassionate care: empowering students through nurse education. Nurse Educ Today. 2014 Sep;34(9):1242-5. doi: 10.1016/j.nedt.2013.07.011. Epub 2013 Jul 25. PMID 23972295
- See also: Compassion care — https://www.aacnnursing.org/5b-tool-kit/themes/compassionate-care